CLINICAL TRIAL: NCT05547451
Title: SARS Cov2 Vaccination in Adolescents From 12 to 18 With Juvenile Idiopathic Arthritis in Angers, Nantes and Rennes : Acceptance and Safety.
Brief Title: SARS Cov 2 Vaccination in Adolescents With Juvenile Idiopathic Arthritis
Acronym: VACOVAJI
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Angers (Other Government); Rennes University Hospital (Other); Clinique de l'Anjou (Other)
Responsible Party: Sponsor
Other Study IDs: RC22_0237
Record Dates: First submitted 2022-09-12; First posted 2022-09-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: SARS Cov 2 Vaccination in Adolescents With Juvenile Idiopathic Arthritis
Keywords: SARS Cov2 vaccination; juvenile idiopathic arthritis; paediatric; safety; acceptance
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial population: Children from 12 to 18 years old followed up for juvenile arthritis in Angers, Nantes and Rennes.

SUMMARY:
Since june 2021, vaccination against the SARS-Cov2 virus is recommanded in France to all children from 12 to 18 years old. In the specific population of teenagers living with juvenile arthritis, the vaccine seems to be safe and well tolerated. It has been shown previously that this population has a vaccine coverage lower than the global population even though few datas are available on this topic The aim of this resarch is to study the vaccination coverage against the SARS-Cov2 virus and more specifically the reasons why adolescents were or were not vaccinated in the population of adolescents with juvenile arthitis followed up in Angers, Nantes and Rennes. For this purpose, a review of the medical record will be done and a questionnaire will be adressed to the family of patients in order to collect informations about the disease, the treatments, the motives or obstacles to vaccination. Secondaries end points are safety of the vaccination, consequences on the juvenile arthritis (such as changes in the medication, flare-up of the illness) and the occurence of covid infection after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 12 to 18 years old, on January the 1st 2022
* Patients followed up from juvenile arthritis
* Patients followed up in 2021 and 2022

Exclusion Criteria:

* Patients under 12 years old.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from 12 to 18 years old followed up from juvenile arthritis in 2021 and 2022 at Angers, Nantes and Rennes.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
SARS Cov2 vaccination coverage of this population and factors influencing the realization of the vaccination. | From june 2021 to December 2022
  Percentage of patients vaccinated

SECONDARY OUTCOMES:
Tolerance of the SARS-Cov2 vaccination | From june 2021 to December 2022
  Occurrence of any side-effects
Effect of the SARS Cov2 vaccination on juvenile arthritis | From june 2021 to December 2022
  Occurrence of flare up of the illness, modification of treatment
SARS-Cov 2 infection after vaccination | From june 2021 to December 2022
  Occurrence and severity of the infection

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided